CLINICAL TRIAL: NCT03159780
Title: Prevalence of Corneal Astigmatism Before Glaucoma Surgery in Chinese Patients With Primary Angle-closure Glaucoma
Status: Completed | Type: Observational
Sponsor: Mingkai Lin (Other)
Responsible Party: Sponsor-Investigator, Mingkai Lin, Head of Glaucoma Center, Zhongshan Ophthalmic Center, Sun Yat-sen University
Organization: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Other Study IDs: ZhongshanOC20170503
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Glaucoma, Angle-Closure; Astigmatism
MeSH Terms: conditions — Glaucoma, Angle-Closure; Astigmatism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clear-lens extraction has been considered as first-line therapy for primary angle closure glaucoma(PACG) and application of toric intraocular lens (IOLs) leads to better postoperative visual acuity, yet little is known about the prevalence of corneal astigmatism in PACG patients. We intend to make biometry examination for Chinese PACG patients, to obtain keratometry (K) , axial length (AL) and so on, and demographics data will also be recorded. We will study the prevalence of corneal astigmatism before glaucoma surgery in Chinese patients with PACG. Furthermore, differences of corneal astigmatism between primary angle-closure glaucoma and cataract patients will be explored. Finally, the prevalence of corneal astigmatism before glaucoma surgery in Chinese patients with PACG will be portrayed and can be instructive to the IOLs' manufactering.

DETAILED DESCRIPTION:
Biometry examination contains keratometry (K) , axial length (AL), central anterior chamber depth, visual field loss(mean deviation, MD), choroidal thickness(CT), range of goniosynechia, and stage of PACG.

Demographics data contains age, gender, and eye.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are phakic and aged 40 years or older , and had newly diagnosed primary angle closure with intraocular pressure 30 mm Hg or greater or primary angle-closure glaucoma, will be recruited during preoperative screening at Zhongshan Ophthalmic Center.

Exclusion Criteria:

* Patients with corneal disease, irregular astigmatism, previous corneal or intraocular surgery, or a history of ocular inflammation will be excluded.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary angle closure was defi ned as iridotrabecular contact, either appositional or synechial, of at least 180° on gonioscopy, and primary angle-closure glaucoma as reproducible glaucomatous visual fi eld defects, glaucomatous optic neuropathy, or both, and intraocular pressure greater than 21 mm Hg on at least one occasion.
Sampling Method: Non-Probability Sample
Enrollment: 808 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of corneal astigmatism | During preoperative screening (1 day)
  Data of corneal astigmatism will be acquired through examination,and different types of corneal astigmatism will be diagnosed and seperated.Moreover,we will analyse the prevalence of corneal astigmatism,and compare among different age groups and different genders.Correlation between demographic features and data will be analysed,too.

SECONDARY OUTCOMES:
Prevalence of keratometry | During preoperative screening (1 day)
  Flat,steep and mean keratometry will be examined before glaucoma surgery. Moreover,we will analyse the prevalence of corneal astigmatism,and compare among different age groups and different genders.
Prevalence of axial length | During preoperative screening (1 day)
  Axial length will be measured by both IOL Master and A-scan, and data will be compared between different measurements,different genders and different age groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mingkai Lin, MD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Azuara-Blanco A, Burr J, Ramsay C, Cooper D, Foster PJ, Friedman DS, Scotland G, Javanbakht M, Cochrane C, Norrie J; EAGLE study group. Effectiveness of early lens extraction for the treatment of primary angle-closure glaucoma (EAGLE): a randomised controlled trial. Lancet. 2016 Oct 1;388(10052):1389-1397. doi: 10.1016/S0140-6736(16)30956-4. PMID 27707497
- [Result] Gao X, Huang W, Wang W, Zhou M, Wang J, Du S, Chen S, Zhang X. Topographic profile of choroid in eyes after acute primary angle-closure. Can J Ophthalmol. 2016 Oct;51(5):354-361. doi: 10.1016/j.jcjo.2016.02.025. Epub 2016 Sep 3. PMID 27769326
- [Result] Chen W, Zuo C, Chen C, Su J, Luo L, Congdon N, Liu Y. Prevalence of corneal astigmatism before cataract surgery in Chinese patients. J Cataract Refract Surg. 2013 Feb;39(2):188-92. doi: 10.1016/j.jcrs.2012.08.060. Epub 2012 Nov 7. PMID 23141077
- [Derived] Zuo C, Gong R, Chen W, Chen C, Su J, Wei K, Gao X, Lin M, Ge J. Investigation of Corneal Astigmatism in Chinese Patients With Primary Angle Closure Disease. J Glaucoma. 2018 Dec;27(12):1131-1135. doi: 10.1097/IJG.0000000000001061. PMID 30134368